CLINICAL TRIAL: NCT01576484
Title: A Phase 2, Open-Label Extension of Study R727-CL-1003 to Evaluate the Long-Term Safety and Efficacy of REGN727 Administered by Subcutaneous Injection in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Open-Label Extension of Study R727-CL-1003 (NCT01266876) to Evaluate the Long-Term Safety and Efficacy of Alirocumab (REGN727) in Participants With Heterozygous Familial Hypercholesterolemia (HeFH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R727-CL-1032
Record Dates: First submitted 2012-03-27; First posted 2012-04-12 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Hypercholesterolemia; Heterozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Matched to Alirocumab (Placebo Comparator): Participants who received placebo in parent study (NCT01576484), has received a subcutaneous injection of placebo matched to alirocumab every 2 weeks for 4 years in this study.
  Interventions: Drug: Placebo Matched to Alirocumab
- Alirocumab 150 mg (Experimental): Participants who received alirocumab in parent study (NCT01576484), has received a subcutaneous injection of alirocumab 150 milligram (mg) every 2 weeks for 4 years in this study.
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Alirocumab — Alirocumab was supplied in a pre-filled syringe and administered subcutaneously (SC) in the abdomen, thigh, or outer upper arm; REGN727(SAR236553) is an anti-PCSK9 (proprotein convertase subtilisin/kexin type 9) antibody
  Other Names: REGN727; SAR236553; PRALUENT
  Arms: Alirocumab 150 mg
Drug: Placebo Matched to Alirocumab — Placebo matched to alirocumab was supplied in a pre-filled syringe and administered subcutaneously (SC) in the abdomen, thigh, or outer upper arm; REGN727(SAR236553) is an anti-PCSK9 (proprotein convertase subtilisin/kexin type 9) antibody
  Arms: Placebo Matched to Alirocumab

SUMMARY:
The primary objective of the study was to assess the long-term safety and tolerability of alirocumab in patients with heFH who were receiving concomitant treatment with hydroxymethyl glutaryl-coenzyme A (HMG-CoA) reductase inhibitors (statins), with or without other lipid-modifying therapies (LMTs).

ELIGIBILITY:
Key Inclusion Criteria:

1. Prior participation in and the successful completion of the R727-CL-1003 study (NCT01266876).
2. Patients must be on a stable daily statin regimen for at least 3 weeks before prior to entry into the study
3. A negative urine pregnancy at the screening/baseline visit for women of childbearing potential

Key Exclusion Criteria:

1. Reported a drug-related serious adverse event (SAE) or drug-related clinical or laboratory adverse event (AE) in the R727-CL-1003 study that resulted in early termination or withdrawal
2. Significant protocol deviation in R727-CL-1003, such as non-compliance by the investigator or patient
3. Low-density lipoprotein (LDL) apheresis within 12 months before the screening/baseline visit

Note: Other exclusion criteria applied

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (14):
- United States (11):
  - Mission Viejo, California
  - Newport Beach, California
  - Thousand Oaks, California
  - Miami, Florida
  - Port Orange, Florida
  - Kansas City, Kansas
  - Auburn, Maine
  - St Louis, Missouri
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Houston, Texas
- Canada (3):
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec

REFERENCES:
- [Derived] Dufour R, Bergeron J, Gaudet D, Weiss R, Hovingh GK, Qing Z, Yang F, Andisik M, Torri A, Pordy R, Gipe DA. Open-label therapy with alirocumab in patients with heterozygous familial hypercholesterolemia: Results from three years of treatment. Int J Cardiol. 2017 Feb 1;228:754-760. doi: 10.1016/j.ijcard.2016.11.046. Epub 2016 Nov 9. PMID 27886619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 sites in the United States and Canada between 28 Feb 2012 and 22 Dec 2016. A total of 59 participants were screened in the study.
Pre-assignment Details: Out of 59, 58 participants received alirocumab in this open-label extension study.
Groups:
- Placebo Participants in Parent Study: Participants who received placebo in parent study (NCT01266876), received a subcutaneous injection of alirocumab 150 milligram (mg) every 2 weeks for 4 years in this study.
- Participants Previously Exposed to Alirocumab in Parent Study: Participants who received alirocumab in parent study (NCT01266876), also received a subcutaneous injection of alirocumab 150 milligram (mg) every 2 weeks for 4 years in this study.
Period: Overall Study
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study
Started | 12 | 46
Completed | 7 | 27
Not Completed | 5 | 19
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Sponsor Decision | 2 | 8
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of 58 patients (46 patients who previously received alirocumab and 12 patients who previously received placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | Total
Number analyzed (Participants) | 12 | 46 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (9.7) | 54.3 (9.4) | 54.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 6 | 32 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 10 | 44 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 11 | 44 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death
Description: An AE was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. Treatment- emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on- treatment period (time from the first dose of study drug to the last dose of study drug plus 70 days). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline (Day 1 of current study) to end of study (Week 218)
Population: Safety Analysis Set (SAF) included all participants who received at least 1 dose or part of a dose of alirocumab.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who received placebo or alirocumab in the parent study (NCT01576484).
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
Participants
  Adverse Events | 12 | 42 | 54
  Serious Adverse Events | 4 | 8 | 12
  Adverse Events Leading to Death | 0 | 0 | 0

2. Secondary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline in the Current Study to Week 24
Description: Percent change for serum LDL-C (Low-density lipoprotein cholesterol) from baseline to Week 24 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) to Week 24
Population: SAF included all participants who received at least 1 dose or part of a dose of alirocumab. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 11 | 44 | 55
percent change | -73.15 (15.01) | -63.40 (22.04) | -65.35 (21.07)

3. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C) From Baseline in Current Study to Week 12
Description: Percent change for serum LDL-C (Low-density lipoprotein cholesterol) from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 44 | 56
percent change | -55.93 (29.53) | -63.94 (23.35) | -62.22 (24.73)

4. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B, Non-High Density Lipoprotein Cholesterol (HDL-C), and Total Cholesterol From Baseline in Current Study to Week 24
Description: Percent change for Apo B, Non-HDL-C and Total Cholesterol from baseline to Week 24 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline(current study) up to Week 24
Population: SAF included all participants who received at least 1 dose or part of a dose of alirocumab. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Apo B: number analyzed (Participants) | 11 | 44 | 55
  Apo B | -52.23 (20.30) | -50.52 (18.18) | -50.86 (18.43)
  Non-HDL-C: number analyzed (Participants) | 12 | 44 | 56
  Non-HDL-C | -56.75 (21.80) | -55.43 (20.97) | -55.71 (20.95)
  Total cholesterol: number analyzed (Participants) | 12 | 44 | 56
  Total cholesterol | -42.72 (15.30) | -41.47 (16.37) | -41.74 (16.02)

5. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B, Non-High Density Lipoprotein Cholesterol (HDL-C), and Total Cholesterol From Baseline in Current Study to Week 12
Description: Percent change for serum Apo B, Non-HDL-C, and Total Cholesterol from baseline to Week 12 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) up to Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Apo- B: number analyzed (Participants) | 11 | 44 | 55
  Apo- B | -40.69 (30.46) | -48.78 (20.24) | -47.16 (22.56)
  Non-HDL- C: number analyzed (Participants) | 12 | 44 | 56
  Non-HDL- C | -47.81 (32.92) | -54.97 (22.85) | -53.44 (25.18)
  Total Cholesterol: number analyzed (Participants) | 12 | 44 | 56
  Total Cholesterol | -36.78 (24.88) | -40.47 (16.93) | -39.68 (18.72)

6. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C) From Baseline in Current Study to Week 52
Description: Percent change for serum LDL-C from baseline to Week 52 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) up to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 42 | 54
percent change | -54.57 (26.20) | -55.67 (34.41) | -55.43 (32.53)

7. Secondary Outcome: Percentage of Participants With Low Density Lipoprotein Cholesterol (LDL-C) Less Than (<) 70 Milligrams Per Deciliter (mg/dL) for Prior Myocardial Infarction (MI)/Stroke, or <100 mg/dL [2.59 mmol/L] for Participants Without Prior MI/Stroke at Week 24
Description: Percentage of participants reaching LDL-C goal (ie, LDL-C <70 mg/dL (1.81 millimoles per liter [mmol/L]) in case of prior MI/stroke, or <100 mg/dL [2.59 mmol/L] for participants without prior MI/stroke) at week 24 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, were reported.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 11 | 44 | 55
Percentage of Participants | 100.00 | 90.91 | 92.73

8. Secondary Outcome: Percent Change in Lipoprotein a (Lp[a]) at Week 24
Description: Percent change in serum lipoprotein a at week 24 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, was reported.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 11 | 44 | 55
percent change | -27.91 (23.62) | -29.41 (25.01) | -29.11 (24.53)

9. Secondary Outcome: Percent Change in High Density Lipoprotein Cholesterol (HDL-C) at Week 24 and Week 12
Description: Percent change for serum High Density Lipoprotein Cholesterol (HDL-C) in the current study at weeks 24 and week 12, during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, was reported.
Time Frame: At Week 24 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Week 24: number analyzed (Participants) | 12 | 44 | 56
  Week 24 | 2.61 (15.75) | 7.14 (16.04) | 6.17 (15.94)
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | 1.46 (14.08) | 10.43 (15.98) | 8.51 (15.91)

10. Secondary Outcome: Percent Change in Lipoprotein a at Week 12
Description: Percent change for serum Lipoprotein a at Week 12 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, was reported.
Time Frame: At Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo Matched to R727: Participants who received placebo in parent study has received a subcutaneous injection of placebo matched to alirocumab every 2 weeks for 4 years in this study.
Arm/Group | Placebo Matched to R727 | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 11 | 44 | 55
percent change | -20.30 (24.10) | -26.98 (22.71) | -25.64 (22.92)

11. Secondary Outcome: Percent Change in Triglycerides (TG) at Week 24 and Week 12
Description: Percent change for serum TG at Week 24 and Week 12 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, was reported.
Time Frame: At Week 24 and 12
Population: SAF included all participants who received at least 1 dose or part of a dose of alirocumab. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Week 24: number analyzed (Participants) | 12 | 44 | 56
  Week 24 | 0.19 (54.71) | -2.01 (41.22) | -1.54 (43.91)
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | -6.40 (46.11) | 0.52 (34.17) | -0.96 (36.69)

12. Secondary Outcome: Percent Change in Apolipoprotein A-1 (Apo A-1) at Week 24 and Week 12
Description: Percent change for serum Apo A-1 at Week 24 and Week 12 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, was reported.
Time Frame: At Week 24 and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Week 24: number analyzed (Participants) | 11 | 44 | 55
  Week 24 | 5.41 (11.96) | 4.78 (11.20) | 4.91 (11.24)
  Week 12: number analyzed (Participants) | 11 | 44 | 55
  Week 12 | 11.10 (11.43) | 8.64 (10.99) | 9.13 (11.02)

13. Secondary Outcome: Percent Change in Low Density Lipoprotein Cholesterol (LDL-C) From Baseline in the Current Study to the End of Treatment
Description: Percent change for serum LDL-C from baseline to Week 208 during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) to the End of Treatment (Week 208)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 3 | 14 | 17
percent change | -52.20 (16.86) | -58.46 (23.51) | -57.36 (22.15)

14. Secondary Outcome: Percentage of Participants With Low Density Lipoprotein Cholesterol (LDL-C) Less Than (<) 70 Milligrams Per Deciliter (mg/dL) for Prior MI/Stroke, or <100 mg/dL [2.59 mmol/L] for Participants Without Prior MI/Stroke at Week 12, 52 and End of Treatment
Description: Percentage of participants reaching LDL-C goal (ie, LDL-C <70 mg/dL (1.81 millimoles per liter [mmol/L]) in case of prior MI/stroke, or <100 mg/dL [2.59 mmol/L] for participants without prior MI/stroke) at week 12, 52 and end of treatment, during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study, were reported.
Time Frame: At Week 12, 52 and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percentage of participants
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | 83.33 | 90.91 | 89.29
  Week 52: number analyzed (Participants) | 12 | 42 | 54
  Week 52 | 75.00 | 83.33 | 81.48
  End of Treatment (Week 208): number analyzed (Participants) | 3 | 14 | 17
  End of Treatment (Week 208) | 100 | 85.71 | 88.24

15. Secondary Outcome: Absolute Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline in the Current Study to Weeks 12, 24, 52, and End of Treatment
Description: Absolute change was reported for serum LDL-C from baseline to weeks 12, 24, 52, and end of Treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) to Weeks 12, 24, 52, and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milligram per Deciliter (mg/dL)
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
Milligram per Deciliter (mg/dL)
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | -92.0 (54.3) | -96.8 (44.7) | -95.8 (46.4)
  Week 24: number analyzed (Participants) | 11 | 44 | 55
  Week 24 | -113.2 (24.9) | -95.3 (40.0) | -98.9 (37.9)
  Week 52: number analyzed (Participants) | 12 | 42 | 54
  Week 52 | -87.0 (44.5) | -83.8 (58.6) | -84.5 (55.4)
  Week 208: number analyzed (Participants) | 3 | 14 | 17
  Week 208 | -80.3 (38.7) | -78.1 (33.6) | -78.5 (33.2)

16. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B, Non-High Density Lipoprotein Cholesterol (HDL-C), Total Cholesterol, Lipoprotein a (Lp[a]), HDL-C, Triglycerides, and Apolipoprotein A-1 From Baseline in Current Study to Week 52 and End of Treatment
Description: Percent change was reported for serum (Apo B), non-HDL-C, total-C, Lp(a), HDL-C, TG, and Apo A-1 from baseline to weeks 52 and end of treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) up to Weeks 52 and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percent change
  Apo B : Week 52: number analyzed (Participants) | 11 | 42 | 53
  Apo B : Week 52 | -43.04 (25.60) | -45.17 (28.51) | -44.73 (27.71)
  Apo B : Week 208: number analyzed (Participants) | 3 | 14 | 17
  Apo B : Week 208 | -45.02 (17.58) | -48.07 (18.61) | -47.53 (17.93)
  Non- HDL-C: Week 52: number analyzed (Participants) | 12 | 42 | 54
  Non- HDL-C: Week 52 | -47.10 (27.26) | -48.60 (31.71) | -48.27 (30.54)
  Non- HDL-C: Week 208: number analyzed (Participants) | 3 | 14 | 17
  Non- HDL-C: Week 208 | -43.29 (17.98) | -50.34 (21.40) | -49.10 (20.50)
  Total -C : Week 52: number analyzed (Participants) | 12 | 42 | 54
  Total -C : Week 52 | -35.09 (19.16) | -36.41 (24.89) | -36.11 (23.57)
  Total -C : Week 208: number analyzed (Participants) | 3 | 14 | 17
  Total -C : Week 208 | -35.33 (11.92) | -37.01 (16.59) | -36.72 (15.55)
  Lp-(a): Week 52: number analyzed (Participants) | 11 | 42 | 53
  Lp-(a): Week 52 | -24.77 (25.14) | -22.91 (30.33) | -23.30 (29.11)
  Lp-(a): Week 208: number analyzed (Participants) | 3 | 14 | 17
  Lp-(a): Week 208 | -23.92 (39.92) | -31.29 (30.20) | -29.99 (30.80)
  HDL-C: Week 52: number analyzed (Participants) | 12 | 42 | 54
  HDL-C: Week 52 | 5.40 (17.64) | 7.74 (14.21) | 7.22 (14.89)
  HDL-C: Week 208: number analyzed (Participants) | 3 | 14 | 17
  HDL-C: Week 208 | -9.83 (12.49) | 4.94 (11.25) | 2.34 (12.49)
  TG : Week 52: number analyzed (Participants) | 12 | 42 | 54
  TG : Week 52 | -6.04 (41.12) | -3.84 (40.25) | -4.33 (40.07)
  TG : Week 208: number analyzed (Participants) | 3 | 14 | 17
  TG : Week 208 | 16.69 (28.93) | -5.28 (23.05) | -1.40 (24.71)
  Apo A-1 : Week 52: number analyzed (Participants) | 11 | 42 | 53
  Apo A-1 : Week 52 | 6.76 (10.82) | 3.90 (10.80) | 4.49 (10.76)
  Apo A-1 : Week 208: number analyzed (Participants) | 3 | 14 | 17
  Apo A-1 : Week 208 | -1.46 (4.48) | 9.53 (7.45) | 7.59 (8.14)

17. Secondary Outcome: Change in Ratio in Apolipoprotein (Apo) B/Apo A-1 From Baseline in Current Study to Week 12, 24, 52, and End of Treatment.
Description: Change in ratio in Apolipoprotein (Apo) B/Apo A-1 from baseline in current Study to week 12, 24, 52, and end of treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: Baseline (current study) to Weeks 12, 24, 52, and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 44 | 56
Ratio
  Change at Week 12: number analyzed (Participants) | 11 | 44 | 56
  Change at Week 12 | -0.397 (0.234) | -0.456 (0.230) | -0.444 (0.230)
  Change at Week 24: number analyzed (Participants) | 11 | 44 | 56
  Change at Week 24 | -0.450 (0.162) | -0.460 (0.211) | -0.458 (0.201)
  Change at Week 52: number analyzed (Participants) | 11 | 42 | 53
  Change at Week 52 | -0.385 (0.210) | -0.416 (0.295) | -0.410 (0.278)
  Change at Week 208: number analyzed (Participants) | 3 | 14 | 17
  Change at Week 208 | -0.330 (0.165) | -0.402 (0.164) | -0.389 (0.161)

18. Secondary Outcome: Percentage of Participants With Apolipoprotein (Apo) B <80 mg/dL at Week 12, 24, 52, and End of Treatment
Description: Percentage of participants was calculated with Apo B <80 mg/dL (0.8 mmol/L) at week 12, 24, 52, and End of Treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: At Week 12, 24, 52, and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percentage of participants
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | 66.67 | 79.55 | 76.79
  Week 24: number analyzed (Participants) | 12 | 44 | 56
  Week 24 | 91.67 | 81.82 | 83.93
  Week 52: number analyzed (Participants) | 12 | 42 | 54
  Week 52 | 66.67 | 73.81 | 72.22
  Week 208: number analyzed (Participants) | 3 | 14 | 17
  Week 208 | 100.00 | 85.71 | 88.24

19. Secondary Outcome: Percentage of Participants With Non-High Density Lipoprotein Cholesterol (HDL-C) <100 mg/dL (2.59 mmol/L) at Week 12, 24, 52, and End of Treatment
Description: Percentage of participants was calculated with non-HDL-C <100 mg/dL (2.59 mmol/L) at Weeks 12, 24, 52, and End of Treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: At Week 12, 24, 52, and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percentage of participants
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | 58.33 | 75.00 | 71.43
  Week 24: number analyzed (Participants) | 12 | 44 | 56
  Week 24 | 91.67 | 81.82 | 83.93
  Week 52: number analyzed (Participants) | 12 | 42 | 54
  Week 52 | 58.33 | 73.81 | 70.37
  Week 208: number analyzed (Participants) | 3 | 14 | 17
  Week 208 | 66.67 | 78.57 | 76.47

20. Secondary Outcome: Percentage of Participants With Low Density Lipoprotein Cholesterol (LDL-C) Less Than (<) 70 Milligrams Per Deciliter (mg/dL) and/or ≥ 50% Reduction in LDL-C (if LDL-C >70 mg/dL [1.81 mmol/L]) at Week 12, 24, 52, and End of Treatment
Description: Percentage of Participants was calculated with LDL-C <70 mg/dL (1.81 mmol/L) and/or ≥ 50% Reduction in LDL-C (if LDL-C >70 mg/dL [1.81 mmol/L]) at Weeks 12, 24, 52, and End of Treatment (Week 208) during the efficacy treatment period, which is defined as the time from the first study drug injection up to 21 days after the last study drug injection in the current study.
Time Frame: At Week 12, 24, 52, and End of Treatment (Week 208)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study | All Participants
Number analyzed (Participants) | 12 | 46 | 58
percentage of participants
  Week 12: number analyzed (Participants) | 12 | 44 | 56
  Week 12 | 66.67 | 86.36 | 82.14
  Week 24: number analyzed (Participants) | 11 | 44 | 55
  Week 24 | 100.00 | 81.82 | 85.45
  Week 52: number analyzed (Participants) | 12 | 42 | 54
  Week 52 | 75.00 | 73.81 | 74.07
  Week 208: number analyzed (Participants) | 3 | 14 | 17
  Week 208 | 66.67 | 85.71 | 82.35

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 218) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events, which are defined as those that are not present at screening, or represent the exacerbation of a pre-existing condition during the treatment period.
Arm/Group | Placebo Participants in Parent Study | Participants Previously Exposed to Alirocumab in Parent Study
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/46
Serious Adverse Events (participants affected / at risk) | 4/12 | 8/46
Other Adverse Events (participants affected / at risk) | 12/12 | 38/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Participants in Parent Study (N=12) | Participants Previously Exposed to Alirocumab in Parent Study (N=46)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Participants in Parent Study (N=12) | Participants Previously Exposed to Alirocumab in Parent Study (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (2)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (8)
Fatigue (General disorders) | 2 (2) | 3 (3)
Injection site bruising (General disorders) | 5 (16) | 6 (10)
Injection site discolouration (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 2 (7) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 7 (10)
Injection site induration (General disorders) | 1 (3) | 0 (0)
Injection site mass (General disorders) | 1 (2) | 2 (5)
Injection site pain (General disorders) | 2 (11) | 4 (5)
Injection site pruritus (General disorders) | 1 (19) | 0 (0)
Injection site swelling (General disorders) | 1 (19) | 1 (1)
Injection site urticaria (General disorders) | 1 (8) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 3 (4)
Bronchitis (Infections and infestations) | 2 (2) | 10 (11)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 3 (5)
Ear infection (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 3 (4)
Influenza (Infections and infestations) | 2 (2) | 5 (5)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 11 (21)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 5 (6)
Tooth infection (Infections and infestations) | 0 (0) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (9) | 13 (22)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (7)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
C-Reactive protein increased (Investigations) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (8) | 8 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (12)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 6 (7)
Headache (Nervous system disorders) | 1 (1) | 10 (12)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (6)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.